CLINICAL TRIAL: NCT01723540
Title: A Comparison of Ultrasonic Dissection Assisted Minilaparotomy Cholecystectomy Versus Laparoscopic Cholecystectomy; a Randomised Two-center Study.
Brief Title: A Comparison of Laparoscopic Cholecystectomy Versus Ultrasonic Dissection Assisted Minilaparotomy Cholecystectomy
Acronym: MC-UsD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5204520
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Postoperative Pain
Keywords: Cholecystectomy,minilaparotomy,laparascopy,ultrasonic dissection
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minilaparotomy cholecystectomy with ultrasonic scissors (Experimental): Minilaparotomy vs laparoscopy
  Interventions: Procedure: Minilaparotomy vs laparoscopy
- Laparoscopic cholecystectomy (Active Comparator): Minilaparotomy vs laparoscopy
  Interventions: Procedure: Minilaparotomy vs laparoscopy

INTERVENTIONS:
Procedure: Minilaparotomy vs laparoscopy — MC-group will undergo ultrasonic dissection assisted minilaparotomy cholecystectomy ans patients in the LC-grout will undergo laparoscopic cholecystectomy

SUMMARY:
Minilaparatomy cholecystectomy with ultrasonic dissection (UsD) is rarely considered and therefore we investigate here the contributions of UsD in early recovery.

ELIGIBILITY:
Inclusion Criteria:- Uncomplicted symptomatic cholelithiasis cholecystitis confirmed by ultrasoud

* ASA physical status 1-3
* Body mass index 18-30
* AGE 18 - 75 years

Exclusion Criteria:

* Pregnancy or lactating
* common bile-duct stones
* acute cholecystitis
* previous upper abdominal operation
* Chirrosis
* Renal disease
* Pancreatitis
* ASA 4-5
* Participation of any other clinical trial within 30 days before the start of the screening period
* History of uncontrolled cardiovascular, epileptic disorder, psychosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Early recovery | One month
  Post operative pain, wound infections, bile leak, mean length of sick leave days, use of analgesics the success of day-surgery

SECONDARY OUTCOMES:
Peroperative outcome | 24 hours
  Operative time, time at the operation theatre, bleeding, length of skin incision

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland